CLINICAL TRIAL: NCT04171869
Title: Towards a Deeper Understanding of Chronic Pediatric Pain: Exploring the Role of Sensory Processing Sensitivity
Brief Title: Survey on Sensory Processing Sensitivity in Chronic Pediatric Pain
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Helen Koechlin, Adjunct senior researcher, University Hospital, Basel, Switzerland
Other Study IDs: Sensory Processing Sensitivity
Record Dates: First submitted 2019-11-14; First posted 2019-11-21 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — observational study, no intervention

SUMMARY:
Background: Pain is defined as an unpleasant sensory and emotional experience and in its chronic form, pain is highly prevalent, up to 25% of children and adolescents are affected by it. The exact etiology of many forms of chronic pain remains unknown. One mechanism that has been proposed to underlie increased pain sensitivity is central sensitization, i.e., increased efficacy of the nervous system in transmitting pain signals, which manifests itself as a lower pain threshold. A lower pain threshold in turn has been recognized as a risk factor for the development of chronic pain. Being more sensitive to pain is one feature commonly shared by those with high sensory processing sensitivity (SPS), who are thought to react more strongly to both positive and negative environmental influences. The relationship between this increased sensitivity and pain tolerance has not been studied to date, but could contribute to our understanding of why some children and adolescents are more vulnerable to developing chronic pain than others.

Objectives and Aims: The aim of this project is to increase scientific understanding of 1) the distribution and correlates of high SPS among children and adolescents suffering from chronic pain, and 2) whether the trait of SPS can help explain increased pain sensitivity and hence vulnerability for chronic pain.

Methods: To determine the distribution (aim 1a) and correlates (aim 1b) of SPS among a population of children and adolescents suffering from chronic pain, an online survey will be conducted. Participants will be asked to complete questionnaires about their SPS as well as pain history and pain characteristics. The distribution of SPS will then be compared to an existing distribution in a sample of healthy children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 17-19 years
* Persistent or recurrent pain for 3 months or more
* Fluent in German or English

Exclusion Criteria:

* Younger than 17 or older than 19 years
* Acute pain

Ages: 17 Years to 19 Years | Sex: All
Age Groups: Child, Adult
Study Population: Adolescents suffering from persistent or recurrent pain for 3 or more months, community sample, recruited mainly via pain clinics
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-05-08 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Highly Sensitive Child Scale | through study completion, an average of 6 months
  Sensory Processing Sensitivity
Functional Disability Inventory for children | through study completion, an average of 6 months
  Physical functioning and disability in children with chronic pain

CONTACTS AND LOCATIONS:
Overall Officials: Helen Koechlin, PhD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Faculty of Psychology, University of Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Yes